CLINICAL TRIAL: NCT05372484
Title: Assessment of New Technologies for the Screening and Diagnosis of Cervical Cancer in Mozambique, A Study to be Conducted in Maputo Central Hospital, Mavalane and Jose Macamo General Hospitals and Mavalane Health Center
Brief Title: Rice Technologies for Cervical Cancer Screening and Diagnosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eduardo Mondlane University (Other); William Marsh Rice University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-0549; NCI-2022-03776 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-25; First posted 2022-05-12 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer
Keywords: Human Papilloma virus; Point-of-care HPV Test; Multimodal Optical Imaging; Screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multi-Modal Optical Imaging (Experimental): Multi-modal imaging (mobile colposcopy and high resolution imaging) of study participants will be performed during the colposcopy examination. Cervical biopsies will be performed using biopsy forceps per standard protocols.
  Interventions: Device: Multimodal optical imaging

INTERVENTIONS:
Device: Multimodal optical imaging — Women referred for colposcopy due to abnormal cervical screening will be recruited into the experimental group of the study. Imaging of study participants will take place during the colposcopy examination.

SUMMARY:
The study aims to compare the accuracy of the lateral flow test to detect HPV at the POC with commercially available HPV test and to determine the diagnostic accuracy and reliability of a multimodal optical imaging system to detect cervical dysplasia, with the gold reference standard of histopathology.

DETAILED DESCRIPTION:
This is a prospective, single-arm community trial involving 678 women aged 25 to 49 years for evaluation of positive cervical cancer screening tests (abnormal cytology, VIA+ and/or HPV+ test). Eligible women will be offered enrollment at the time of their consultation for a follow-up of their abnormal cervical cancer screening test.

Participating centers include: 1) Mavalane Hospital and Health Center and 2) José Macamo General Hospital (José Macamo), 3) Maputo Central Hospital. After providing the informed consent, the participant will answer a short questionnaire that will include demographic information and medical background, including HIV status (HIV-negative, positive, or unknown, and, among women with HIV-positive tests, HIV viral load and CD4 cell count, if available), and cervical cancer screening test results.

The patient will undergo a rapid urine - POC pregnancy test (within 14 days from the date of enrollment). Each participant will then receive instructions and will provide two cervico-vaginal samples taken by the patient herself (self-collection).

The patient will then undergo a pelvic examination with two cervical samples taken by the healthcare provider. 7. A sample taken by the patient herself (self-collection) and a sample taken by the provider will be sent for an HPV test using GeneXpert. Similarly, samples taken by the patient herself (self-collection) and collected by the provider will be stored for the Rice POC rapid HPV test.

The patient will then undergo multimodal imaging. Images/videos of the cervix will be obtained using the mobile colposcope/smartphone and HRME images/videos will be also obtained.

ELIGIBILITY:
Inclusion Criteria:

1. 25 - 49 year old women
2. Women with a positive cervical cancer screening test (abnormal cytology, positive VIA and/or positive HPV test)
3. Women with intact cervix
4. Women who are not pregnant and with a negative pregnancy test (within 14 days from the date of enrollment) ) and not currently breastfeeding
5. Willing and capable of providing informed consent

Exclusion Criteria:

1. Women under 25 or over 49 years old
2. Women who have undergone a total hysterectomy (with removal of the cervix)
3. Women who are pregnant or breastfeeding

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 678 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Development of multimodal optical imaging system | through study completion, an average of 1 year
  Image data will be used as a training set to develop and refine image analysis algorithms. Multimodal Mobile Colposcope will be compared with colposcopic impression considering clinical performance (sensitivity, specificity, positive and negative predictive values, and area under the Receiver Operating Characteristic (ROC) curve)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Schmeler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- M D Anderson Cancer Center, Houston, Texas, United States
- Mozambique (3):
  - José Macamo General Hospital and Health Center, Maputo
  - Maputo Central Hospital, Maputo
  - Mavalane Hospital and Health Center, Maputo

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org